CLINICAL TRIAL: NCT06441617
Title: Confirmatory Trial for Alleviating Fatigue in Multiple Sclerosis
Acronym: CAFE-MS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Accelerated Cure Project for Multiple Sclerosis (Other)
Collaborators: Congressionally Directed Medical Research Programs (U.S. Federal Agency); United States Department of Defense (U.S. Federal Agency); Charite University, Berlin, Germany (Other); University Medical Center Goettingen (Other); US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ACP-CAFE-MS-001; CDMRP- MS220136 (Other Grant/Funding Number: Congressionally Directed Medical Research Programs (CDMRP))
Record Dates: First submitted 2024-05-29; First posted 2024-06-04 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Multiple Sclerosis; Fatigue
MeSH Terms: conditions — Multiple Sclerosis; Fatigue

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be blinded with respect to Program A and Program B. However, the third arm of the trial, Treatment as Usual, will not be blinded. Since outcome assessments are collected online via surveys, the outcome assessor is a blinded entity.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Fatigue Program A added to Treatment as Usual (Experimental): An MS-specific fatigue management program, delivered as a stand-alone, fully automated intervention via an internet-browser.
  Interventions: Device: Online Program for Fatigue
- Fatigue Program B added to Treatment as Usual (Active Comparator): Fatigue Program B will use a web-based interface with similar design and functionality as Fatigue Program A.
  Interventions: Device: Online Program for Fatigue
- Treatment as Usual (No Intervention)

INTERVENTIONS:
Device: Online Program for Fatigue — An MS-specific fatigue management program, delivered as a stand-alone, fully automated intervention via an internet-browser.
  Arms: Fatigue Program A added to Treatment as Usual; Fatigue Program B added to Treatment as Usual

SUMMARY:
CAFE-MS will assess the effectiveness of two online programs for fatigue in multiple sclerosis (MS). Although they differ, both of these online programs contain information about MS and fatigue intended to help people with MS understand and manage their fatigue.

This large-scale, decentralized clinical trial is projected to enroll 2,000 people with MS. The collaboration between iConquerMS and 5 Veterans Affairs (VA) sites in the MS Centers of Excellence is designed to ensure sufficient representation of people with MS from populations traditionally under-represented in MS clinical trials.

The study is a 3-arm, randomized controlled clinical trial with study participation lasting 1 year. Two of the trial arms will include one of two online programs for managing fatigue in MS added to the trial participants' usual MS treatment, and the third arm will include usual MS treatment alone. The online program phase of the trial lasts for 6 months after randomization followed by a final study visit at 12 months. Participants in the usual MS treatment alone arm for the first 6 months will have an opportunity to choose one of the online programs for the final 6 months of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent by person with MS
* Living in the US
* Age ≥ 22
* Confirmed diagnosis of MS by a physician, who is a neurologist or has access to a neurologist's statement of diagnosis
* Fatigue Severity Scale score at or above eligibility threshold
* Fluent in English
* Willingness to engage in self-administration of an online intervention for 24 weeks and complete follow-up assessments
* Access to the internet and e-mail with a compatible device (smartphone, computer, or tablet)
* No MS relapse / no steroid treatment in the 4 weeks prior to answering the screening questionnaire (self-reported)
* No disease-modifying therapeutic (DMT) started in the 4 weeks prior to answering the screening questionnaire (self-reported)

Exclusion Criteria:

* Unwilling or unable to consent
* Refusal to saving, processing and forwarding of pseudonymized data
* Concurrent participation in another interventional trial

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2024-12-05 (Actual); Primary Completion 2027-02-15 (Estimated); Study Completion 2027-09-14 (Estimated)

PRIMARY OUTCOMES:
Chalder Fatigue Scale | Day 180
  The scale contains 11 items covering physical fatigue (items 1-7) and mental fatigue (items 8-11).

SECONDARY OUTCOMES:
PROMIS FatigueMS-8a | Day 180
  The PROMIS FatigueMS-8a questionnaire has eight 5-point Likert scale items on different aspects of fatigue.
PROMIS MS Health | Day 180
  PROMIS MS Health has 14 domains, each comprising four 5-point Likert scale items, covering mobility limitations, spasticity, reduced hand and arm function, fatigue, pain, numbness, cognition issues, sleep disturbances, bowel and bladder dysfunction, vision problems, dizziness and vertigo, sexual dysfunction, mood and emotional changes plus a single 5-point Likert scale item for overall health.
SymptoMScreen | Day 180
  SymptoMScreen has twelve 7-point Likert scale items covering how each of the following MS symptoms affects everyday life activities: walking, hand function, spasticity, pain, sensory function, bladder control, fatigue, vision, dizziness, cognitive function, depression and anxiety.
Frenchay Activities Index | Day 180
  The Frenchay Activities Index (FAI) is a measure of instrumental activities of daily living (IADL) for use with patients with neurological disorders. The FAI assesses a broad range of activities associated with everyday life that the patient has participated in within the recent past, broken into 3 domains: domestic chores, leisure/work, and outdoor activities.

OTHER OUTCOMES:
Treatment Acceptability | Day 180
  The Treatment Acceptability questionnaire consists of seven 5-point Likert items covering affective attitude, burden, ethicality, intervention coherence, opportunity costs, perceived effectiveness, and self-efficacy.

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Washington VA Medical Center, Washington D.C., District of Columbia
  - Baltimore VA Medical Center, Baltimore, Maryland
  - iConquerMS, Waltham, Massachusetts
  - Portland VA Medical Center, Portland, Oregon
  - Nashville VA Medical Center, Nashville, Tennessee
  - Seattle VA Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided